CLINICAL TRIAL: NCT06849479
Title: Effect of Aerobic Exercises on Persisted Post Burn Anemia
Brief Title: Aerobic Exercises on Persisted Post Burn Anemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira saad mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.Rec/012/005217
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group includes 20 patients who had severe burn with total body surface area ranged from 20% to 35%. These patients will receive aerobic exercises in addition to medical treatment of anemia.
  Interventions: Procedure: Aerobic exercise and medical treatment; Dietary Supplement: Medical treatment group
- Group B (Placebo Comparator): This group includes 20 patients who had severe burn with total body surface area ranged from 20 to 35%. These patients will receive a medical treatment of anemia.
  Interventions: Dietary Supplement: Medical treatment group

INTERVENTIONS:
Procedure: Aerobic exercise and medical treatment — Aerobic exercise training was done for 30 minutes, day after day (3 sessions weekly) for 6 weeks. Each session started by warming up phase that was walking on treadmill for 5 minutes at 20% of target heart rate. Active phase after warming up was walking on treadmill for 20 min at 50-70 % of target heart rate. And cooling down phase after the active phase of exercise was walking on treadmill for 5 minutes at 20 % of the target heart rate
  Arms: Group A
Dietary Supplement: Medical treatment group — patient received supplement in the form of one capsule daily, that contain iron supplement (10 mg) and multi vitamins (B1=0.6 mg;, B2=0.6 mg; B6=0.6 mg; B12= 1.2 mc and C=30 mg) as well as essential trace elements (Zinc=5 mg; Copper=0.44 mg; Folic acid=200 mc and Biotin=12 mc

SUMMARY:
Fourty patients who have total body surface area ranged from 20% to 35% of burn, anemic and 8th to 16th week post burn will participate in this study, the patients will be randomly divided into two equal groups (20 patients for each group): Group A (Experimental Group) (Aerobic exercise and medical treatment):

Group B ( Control Group) (Medical treatment group):

ELIGIBILITY:
Inclusion Criteria:

The subject selection will be according to the following criteria:

1. Ages of patients will be ranged from 20 to 35 years.
2. All patients underwent severe burn with TBSA ranged from 20% to 35%.
3. 8 th to 16th week post burn.
4. All patients will be referred with persisted anemia by a surgeon before starting the study procedure.
5. All patients will enter the study having their informed consent

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria: 16

1. Patients with persisted pre burn anemia associated with systematic chronic disease such as coronary artery disease or chronic kidney disease.
2. Patients with pre burn persisted anemia associated with autoimmune disease such as Rheumatoid arthritis, Systemic lupus erythematosus ,Vasculitis, Sarcoidosis, Inflammatory bowel disease (IBD).
3. Unevaluated cardiac arrhythmia, Chronic bronchitis, poorly controlled type 1 diabetes, Extreme morbid obesity, Extreme underweight body mass index less than 12, Poorly controlled hypertension, Poorly controlled seizure disorder, Poorly controlled hyperthyroidism, Orthopedic limitation as fracture, .

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Red blood cells | pre intervention and re assessed after 6 weeks of treatment
  It will be drawn by the doctor and a specialist nurse. Red blood cell (RBC) count measures the number of red blood cells in your blood. The unit of measurements is cell per microliter.
  Normal RBC ranges are: Male: 4.7 to 6.1 million cells per microliter (cells/mcL) Female: 4.2 to 5.4 million cells/mcL.
Hemoglobin | pre intervention and re assessed after 6 weeks of treatment
  It will be drawn by the doctor and a specialist nurse. The unit of measurement is grams/deciliter.
  Normal range for men is , 13.2 to 16.6 grams per deciliter. Normal range for women is, 11.6 to 15 grams per deciliter.
Hematocrit | pre intervention and re assessed after 6 weeks of treatment
  It will be drawn by the doctor and a specialist nurse. The hematocrit is the percentage of packed RBCs in the whole blood. The hematocrit has the implied units of L/L, although it is usually reported as a percent.
  Normal range for Males: 41% to 50%. Normal range for Females: 36% to 44%.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt